CLINICAL TRIAL: NCT06885060
Title: Exploring Eye Vergence Markers in Attention Deficit Hyperactivity Disorder (ADHD) and Autism Spectrum Disorder (ASD).
Brief Title: Exploring Eye Vergence Markers ADHD) and ASD
Status: Active, not recruiting | Type: Observational
Sponsor: Elizabeth Kilbey (Other)
Collaborators: Braingaze (Industry)
Responsible Party: Sponsor-Investigator, Elizabeth Kilbey, Consultant Clinical Psychologist, Child And Adult Neurodevelopment Assessment Ltd
Organization: Child And Adult Neurodevelopment Assessment Ltd (Other)
Other Study IDs: 347961
Record Dates: First submitted 2025-03-07; First posted 2025-03-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD); Autism Spectrum Disorder (ASD)
Keywords: ADHD; ASD; Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorder; Autism; Inattention; Impulsivity; Eye Vergence; Eye Tracking; Hyperactivity; Cognitive Eye Vergence; BGaze Clinic; Bio-marker
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder; Autistic Disorder; Impulsive Behavior; Spasm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ADHD Group: Patients who have a diagnosis of ADHD (but not ASD), either prior to, or diagnosed during, the duration of their participation in the study.
  Interventions: Device: BGaze ADHD Diagnostic Test; Device: Oddball/Alerting Computer Task; Device: Facical Emotion Computer Task
- ASD Group: Patients who have a diagnosis of ASD (but not ADHD), either prior to, or diagnosed during, the duration of their participation in the study.
  Interventions: Device: BGaze ADHD Diagnostic Test; Device: Oddball/Alerting Computer Task; Device: Facical Emotion Computer Task
- Combined Group: Patients who have a combined diagnosis of ADHD and ASD, either prior to, or diagnosed during, the duration of their participation in the study.
  Interventions: Device: BGaze ADHD Diagnostic Test; Device: Oddball/Alerting Computer Task; Device: Facical Emotion Computer Task
- Control Group: Patients who do not have a diagnosis of neither ADHD and/or ASD, and do not show traits of either diagnosis.
  Interventions: Device: BGaze ADHD Diagnostic Test; Device: Oddball/Alerting Computer Task; Device: Facical Emotion Computer Task

INTERVENTIONS:
Device: BGaze ADHD Diagnostic Test — The BGaze Clinic ADHD diagnostic test will be administered to all participants. This involves a computer-based task, where an eye-tracker will be recording their eye-movements.
Device: Oddball/Alerting Computer Task — Oddball/Alerting Computer Task will be completed by all participants while an eye-tracker records their eye movements.
Device: Facical Emotion Computer Task — The Facial Emotion Computer Task will also be completed by all participants while their eye movements are recorded using an eye-tracker.

SUMMARY:
The investigators study aims to evaluate the utility of eye vergence, an eye-tracking measure, as an indicator of visuo-spatial attention in children aged 4-17 years and adults, using computer-based eye-tracking tasks. Eye vergence, a binocular movement crucial for depth perception, has recently been linked to attentional control and neurodevelopmental conditions (NDCs) like ADHD and ASD. The investigators will work with children and adults from the CAN and Beckenham clinical centres to explore the relationship between eye vergence and diagnostic categories, potentially identifying subgroups with specific or overlapping attentional differences. This research may aid in the early detection of attention deficits, informing targeted treatments.

The investigators will compare neuropsychological and behavioural data from routine clinical sessions with neurophysiological data collected via eye-tracking in a large sample of children aged 7-17 and adults with ADHD and ASD. These clinical measures are well-validated. The study will assess the modulation of eye vergence, pupil size, and head movements across tasks that target different attentional processes, such as orienting, disengaging, inhibiting, and sustaining attention. These tasks will be adapted from both Braingaze's battery and other validated eye-tracking tasks.

Additionally, the investigators will explore whether AI can enhance the accuracy of rating scales and questionnaires used to measure ADHD and ASD symptoms in children and adults. With consent, the investigators will use data from previously diagnosed patients collected during routine assessments at the CAN and Beckenham centres.

The investigators will also test the accuracy of using a smartphone selfie camera as an eye tracker. In a subset of 50 children (25 clinical and 25 controls), the investigators will evaluate this technology for its ability to measure eye vergence and identify attentional differences.

This study qualifies as basic science because it aims to explore fundamental mechanisms of eye vergence and its relationship with attention, rather than evaluating or marketing a medical device for diagnosis or treatment. The primary objective is to understand how eye vergence, as a neurophysiological measure, correlates with attentional processes in individuals with ADHD and ASD. Although the study utilizes an eye-tracking device, it does so as a research tool to collect data on visual and cognitive processes. The focus is on expanding the knowledge of cognitive function and attention regulation in neurodevelopmental conditions, not on testing or validating the device for clinical use. This distinction makes the study appropriate for review by the receiving REC as basic scientific research, rather than as a clinical trial of a medical device.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Groups: Patients currently undergoing or who have previously undergone an assessment for either ADHD and/or Autism at either the CAN centre or Dr Kilbey's private practice in Beckenham.
* Control Group: Subjects without a diagnosis of either ADHD nor Autism, who show no traits of these conditions.
* People of any gender/sex who are aged older than 6 years old.

Exclusion Criteria:

* Those with non-corrected vision - e.g. near-sightedness, far-sightedness, strabismus or nystagmus
* Individuals with any other oculomotor deficiency, blindness or vision loss.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals from the Southeast of England, who are able to travel to either New Malden or Beckenham to partake in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the sensitivity and specificity of cognitive eye vergence data, gathered using eye-tracking, for correctly identifying specific attentional deficits in patients with NDCs such as ADHD and ASD. | From enrollment of the first participant, through to study completion after 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Hans A Super, BSc MSc PhD, Study Director — Braingaze & University of Barcelona
Locations (3):
- Braingaze SL, Barcelona, Catalonia, Spain
- United Kingdom (2):
  - The Dr Kilbey Practice, Beckenham, London
  - Child and Adult Neurodevelopment Assessment Ltd, New Malden, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romeo A, Leonovych O, Sole Puig M, Super H. Cognitive Vergence Recorded with a Webcam-Based Eye-Tracker during an Oddball Task in an Elderly Population. Sensors (Basel). 2024 Jan 30;24(3):888. doi: 10.3390/s24030888. PMID 38339605
- [Background] Hashemi, A. et al. (2023) 'Classification of MCI patients using vergence eye movements and pupil responses obtained during a visual oddball test', Aging and Health Research, 3(1), p. 100121. Available at: https://doi.org/10.1016/j.ahr.2023.100121
- [Background] Bast N, Boxhoorn S, Super H, Helfer B, Polzer L, Klein C, Cholemkery H, Freitag CM. Atypical Arousal Regulation in Children With Autism but Not With Attention-Deficit/Hyperactivity Disorder as Indicated by Pupillometric Measures of Locus Coeruleus Activity. Biol Psychiatry Cogn Neurosci Neuroimaging. 2023 Jan;8(1):11-20. doi: 10.1016/j.bpsc.2021.04.010. Epub 2021 Apr 27. PMID 33930603
- [Background] Bustos-Valenzuela, P. et al. (2022) 'Atypical cognitive vergence responses in children with attention deficit hyperactivity disorder but not with autism spectrum disorder in a facial emotion recognition task', Psychiatry Research Communications, 2(2), p. 100045. Available at: https://doi.org/10.1016/j.psycom.2022.100045
- [Background] Jimenez EC, Sierra-Marcos A, Romeo A, Hashemi A, Leonovych O, Bustos Valenzuela P, Sole Puig M, Super H. Altered Vergence Eye Movements and Pupil Response of Patients with Alzheimer's Disease and Mild Cognitive Impairment During an Oddball Task. J Alzheimers Dis. 2021;82(1):421-433. doi: 10.3233/JAD-201301. PMID 34024820
- [Background] Jimenez EC, Avella-Garcia C, Kustow J, Cubbin S, Corrales M, Richarte V, Esposito FL, Morata I, Perera A, Varela P, Canete J, Faraone SV, Super H, Ramos-Quiroga JA. Eye Vergence Responses During an Attention Task in Adults With ADHD and Clinical Controls. J Atten Disord. 2021 Jul;25(9):1302-1310. doi: 10.1177/1087054719897806. Epub 2020 Jan 20. PMID 31959011
- [Background] Sole Puig M, Romeo A, Super H. Vergence eye movements during figure-ground perception. Conscious Cogn. 2021 Jul;92:103138. doi: 10.1016/j.concog.2021.103138. Epub 2021 May 19. PMID 34022640
- [Background] Jimenez EC, Romeo A, Perez Zapata L, Sole Puig M, Bustos-Valenzuela P, Canete J, Varela Casal P, Super H. Eye vergence responses in children with and without reading difficulties during a word detection task. Vision Res. 2020 Apr;169:6-11. doi: 10.1016/j.visres.2020.02.001. Epub 2020 Mar 3. PMID 32143068
- [Background] Boxhoorn S, Bast N, Super H, Polzer L, Cholemkery H, Freitag CM. Pupil dilation during visuospatial orienting differentiates between autism spectrum disorder and attention-deficit/hyperactivity disorder. J Child Psychol Psychiatry. 2020 May;61(5):614-624. doi: 10.1111/jcpp.13179. Epub 2019 Dec 18. PMID 31853987
- [Background] Esposito FL, Super H. Eye vergence responses to novel and familiar stimuli in young children. Acta Psychol (Amst). 2019 Feb;193:190-196. doi: 10.1016/j.actpsy.2019.01.007. Epub 2019 Jan 15. PMID 30654274
- [Background] Esposito FL, Super H. Vergence responses to face stimuli in young children. Neuroreport. 2018 Feb 7;29(3):219-223. doi: 10.1097/WNR.0000000000000963. PMID 29324520
- [Background] Super, H. et al. (2017) 'Neurobiological marker for child and adult ADHD diagnoses', European Psychiatry, 41(S1), pp. S454-S455. Available at: https://doi:10.1016/j.eurpsy.2017.01.489
- [Background] Sole Puig M, Romeo A, Canete Crespillo J, Super H. Eye vergence responses during a visual memory task. Neuroreport. 2017 Feb 8;28(3):123-127. doi: 10.1097/WNR.0000000000000734. PMID 28121809
- [Background] Sole Puig M, Pallares JM, Perez Zapata L, Puigcerver L, Canete J, Super H. Attentional Selection Accompanied by Eye Vergence as Revealed by Event-Related Brain Potentials. PLoS One. 2016 Dec 14;11(12):e0167646. doi: 10.1371/journal.pone.0167646. eCollection 2016. PMID 27973591
- [Background] Sole Puig M, Perez Zapata L, Puigcerver L, Esperalba Iglesias N, Sanchez Garcia C, Romeo A, Canete Crespillo J, Super H. Attention-Related Eye Vergence Measured in Children with Attention Deficit Hyperactivity Disorder. PLoS One. 2015 Dec 22;10(12):e0145281. doi: 10.1371/journal.pone.0145281. eCollection 2015. PMID 26694162
- [Background] Sole Puig M, Puigcerver L, Aznar-Casanova JA, Super H. Difference in visual processing assessed by eye vergence movements. PLoS One. 2013 Sep 19;8(9):e72041. doi: 10.1371/journal.pone.0072041. eCollection 2013. PMID 24069140
- [Background] Sole Puig M, Perez Zapata L, Aznar-Casanova JA, Super H. A role of eye vergence in covert attention. PLoS One. 2013;8(1):e52955. doi: 10.1371/journal.pone.0052955. Epub 2013 Jan 31. PMID 23382827
- See also: Braingaze Website — https://braingaze.com/
- See also: CAN Website — https://www.cancentre.co.uk/
- See also: The Dr Kilbey Practice Website — http://www.drkilbey.com/